CLINICAL TRIAL: NCT00696254
Title: Impact of General Anaesthetics on Excitability of the Peripheral Sensory Nerve
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Other Study IDs: 5-2008
Record Dates: First submitted 2008-03-17; First posted 2008-06-12 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Scheduled for Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: Nerve excitability measurement

SUMMARY:
The aim of this study is to investigate the effect of general anaesthetics on nerve excitability. We use the method of threshold tracking to measure selected parameters of nerve excitability.

ELIGIBILITY:
Inclusion criteria: German speaking patients scheduled for surgery under general anaesthesia.

Weight 50 - 100 kg signed informed consent

Exclusion criteria: 1. known peripheral neuropathy 2. Diabetes mellitus 3. Neuro-psychiatric Diagnosis 4. pregnant/ breast-feeding women 5. congestive heart disease 6. more than 2 risk factors (out of 4) for PONV (female, non-smoker, known PONV, opioids postoperatively) 7. participants of other studies 8. inability of verbal expression

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria: German speaking patients scheduled for surgery under general anaesthesia
Sampling Method: Non-Probability Sample
Dates: Start 2008-03; Study Completion 2008-12

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland